CLINICAL TRIAL: NCT00661687
Title: A Study to Evaluate the Product Performance of the Redesigned Bausch & Lomb PureVision® Contact Lens (Test) Compared to the Currently Marketed Bausch & Lomb PureVision® Contact Lens (Control) When Worn on an Extended Wear Basis.
Brief Title: Comparative Performance of PureVision Lens Designs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 544
Record Dates: First submitted 2008-04-16; First posted 2008-04-18 (Estimated); Results first posted 2010-10-15 (Estimated); Last update posted 2011-12-12 (Estimated); Status verified 2011-12

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Purevision Contact Lens #1 (Active Comparator): PureVision Soft Contact Lens Design (currently marketed)
  Interventions: Device: Currently Marketed PureVision Contact Lens.
- PureVision Contact Lens #2 (Experimental): Redesign of the currently marketed PureVision soft contact lens.
  Interventions: Device: Alternate Design of the PureVision Contact Lens.

INTERVENTIONS:
Device: Currently Marketed PureVision Contact Lens. — Contact lens for continuous wear
  Arms: Purevision Contact Lens #1
Device: Alternate Design of the PureVision Contact Lens. — Contact lens for continuous wear
  Arms: PureVision Contact Lens #2

SUMMARY:
The objective of this study is to evaluate the performance of the PureVision Lens designs when worn on a 30-day continuous wear basis

ELIGIBILITY:
Inclusion Criteria:

* subject is myopic
* VA correctable to 0.3 logMAR or better (driving vision)
* Clear central cornea

Exclusion Criteria:

* Systemic disease affecting ocular health
* using systemic or topical medications
* wear monovision, multifocal or toric contact lenses
* Any grade 2 or greater slit lamp findings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2007-12; Primary Completion 2008-02 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Cairns, MCOptom, PhD, Study Director — Bausch & Lomb Incorporated; Benny Chian, MCOptom, Principal Investigator — Laser Focus Sdn Bhd, Vision Correction Centre; Harvey Siy Uy, MD, Principal Investigator — Asian Eye Institute
Locations (2):
- Laser Focus Sdn Bhd, Vision Correction Centre, Johor Bahru, Johor Bahru, Malaysia
- Asian Eye Institute, Makati City, Philippines

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began on 12/24/07 and lasted for 1 month. Participants were recruited from 10 Asian Sites.
Pre-assignment Details: 206 participants were enrolled. 204 participants were eligible and 189 completed the study. Study was a contralateral design with one eye of each patient randomly assigned to the experimental group and fellow eye to the control group.
Groups:
- PureVision Contact Lens: PureVision Contact Lens, Original Design and Alternate Design. Subjects randomly assigned to receive the Purevision test lens in one eye and the marketed Purevision lens in the fellow eye.
Period: Overall Study
Arm/Group | PureVision Contact Lens
Started | 204 (Contralateral study design, numbers indicate number of subjects.)
Completed | 189 (Number indicates number of subjects successfully completing study.)
Not Completed | 15
Not completed — Study related symptoms and complaints | 5
Not completed — Positive slit lamp findings | 4
Not completed — Inability to maintain wearing schedule | 3
Not completed — Physician Decision | 1
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Groups:
- PureVision Contact Lens: PureVision Contact Lens Original Design and New Design.
Arm/Group | PureVision Contact Lens
Number analyzed (Participants) | 204
Age Continuous [Mean (Standard Deviation); unit: Years] — Mean and standard deviation measured on the eligible population of 204
  Years | 28.1 (6.97)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender was measured in the eligible population of 204 participants (408 eyes).
  Participants
    Female | 130
    Male | 74
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 203
  White | 1

OUTCOME MEASURES:

1. Primary Outcome: Subjective Responses to Symptoms/Complaints
Description: Subjective responses to symptoms/complaints on a scale 0-100, where 100 is the most favorable score. Subjects rated various aspects of lens comfort, vision, and handling. The average of each symptom/complaint over all follow-up visits was assessed as the primary endpoint.
Time Frame: Measured at screening/dispensing visit, 1 day, 1 week and 1 month follow-up visits
Population: All eligible participants
Measure: Mean (Standard Deviation); unit: Visual Analogue Scale
Units Other Than Participants: eyes
Groups:
- PureVision Contact Lens Design #1: PureVision soft contact lens (currently marketed).
- PureVision Contact Lens Design #2: Redesign of the currently marketed PureVision soft contact lens.
Arm/Group | PureVision Contact Lens Design #1 | PureVision Contact Lens Design #2
Number analyzed (Participants) | 102 | 102
Number analyzed (eyes) | 204 | 204
Visual Analogue Scale | 80.0 (15.07) | 81.2 (14.52)

2. Secondary Outcome: LogMAR Visual Acuity
Description: The mean distance high contrast LogMAR visual acuity (VA) score for test eyes over all visits, determined by the total number of letters correctly identified on the logMAR chart.
Time Frame: Mean over all visits - 1 day, 1 week, 1 month
Population: All Eligible, Dispensed Eyes
Measure: Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: eyes
Arm/Group | PureVision Contact Lens Design #1 | PureVision Contact Lens Design #2
Number analyzed (Participants) | 102 | 102
Number analyzed (eyes) | 204 | 204
LogMAR | 0.001 (0.0678) | 0.003 (0.0673)

3. Secondary Outcome: Lens Characteristics
Description: Investigators evaluated study lenses, while on eye, for the number of eyes showing 100% wettability, no discoloration, none-light deposits, fully centered centration, and adequate movement.
Time Frame: Over all scheduled visits day 1 - 1 month
Population: Over All Scheduled Visits, All Eligible, Dispensed Eyes
Measure: Number; unit: Eyes
Units Other Than Participants: eyes
Arm/Group | PureVision Contact Lens Design #1 | PureVision Contact Lens Design #2
Number analyzed (Participants) | 102 | 102
Number analyzed (eyes) | 204 | 204
Eyes
  Lens wettability - 100% of anterior surface | 75 | 78
  Lens discoloration - absent | 182 | 182
  Suboptimal lens deposits (medium/heavy) - absent | 181 | 179
  Lens centration - excellent | 171 | 164
  Lens movement - adequate | 138 | 138

ADVERSE EVENTS:
Time Frame: 1 month
Groups:
- PureVision Contact Lens Design #1: PureVision Contact Lens, Original Design. Subjects randomly assigned to receive the Purevision test lens in one eye and the marketed Purevision lens in the fellow eye.
- PureVision Contact Lens Design #2: PureVision Contact Lens Test Design. Subjects randomly assigned to receive the Purevision test lens in one eye and the marketed Purevision lens in the fellow eye
Arm/Group | PureVision Contact Lens Design #1 | PureVision Contact Lens Design #2
Serious Adverse Events (participants affected / at risk) | 0/204 | 0/204
Other Adverse Events (participants affected / at risk) | 0/204 | 0/204

LIMITATIONS AND CAVEATS:
2 participants discontinued due to adverse events, not classified as serious. One subject in the test group developed corneal ulcer, one subject in the control group developed a central epithelial defect, both conditions resolved following treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less